CLINICAL TRIAL: NCT00703261
Title: A Randomized, Double-Blind, Parallel Group Study to Evaluate the Effects of High Dose Statin Therapy on 18Fluorine Fluorodeoxyglucose (18FDG) Uptake in Arteries of Patients With Atherosclerotic Vascular Disease
Brief Title: Evaluate the Utility of 18FDG-PET as a Tool to Quantify Atherosclerotic Plaque (MK-0000-081 AM3)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-081; 2007_651
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Results first posted 2011-11-30 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Atherosclerotic Vascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 10 mg Atorvastatin (Active Comparator): 10 mg atorvastatin + placebo
  Interventions: Drug: atorvastatin; Drug: placebo
- 80 mg Atorvastatin (Active Comparator): 80 mg atorvastatin + placebo
  Interventions: Drug: atorvastatin; Drug: placebo

INTERVENTIONS:
Drug: atorvastatin — Participants will be asked to self-administer one atorvastatin 10 mg or 80 mg tablet at approximately the same time each day.
  Other Names: Lipitor
Drug: placebo — Participants will be asked to self-administer one tablet of placebo to atorvastatin 10 mg or 80 mg at approximately the same time each day.

SUMMARY:
The purpose of this study is to evaluate the utility of 18Fluorine Fluorodeoxyglucose Positron Emission Tomography (18FDG-PET) as a tool to quantify atherosclerotic plaque.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ages 30 to 80
* Participant is on a low dose statin for at least 6 weeks prior to screening or is statin-naive at screening

Exclusion Criteria:

* Participant has human immunodeficiency virus (HIV), Hepatitis B or C
* Participant uses illegal drugs
* Participant has Type I diabetes
* Participant has a history of claustrophobia

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Singh P, Emami H, Subramanian S, Maurovich-Horvat P, Marincheva-Savcheva G, Medina HM, Abdelbaky A, Alon A, Shankar SS, Rudd JH, Fayad ZA, Hoffmann U, Tawakol A. Coronary Plaque Morphology and the Anti-Inflammatory Impact of Atorvastatin: A Multicenter 18F-Fluorodeoxyglucose Positron Emission Tomographic/Computed Tomographic Study. Circ Cardiovasc Imaging. 2016 Dec;9(12):e004195. doi: 10.1161/CIRCIMAGING.115.004195. PMID 27956407
- [Derived] Subramanian S, Emami H, Vucic E, Singh P, Vijayakumar J, Fifer KM, Alon A, Shankar SS, Farkouh M, Rudd JHF, Fayad ZA, Van Dyke TE, Tawakol A. High-dose atorvastatin reduces periodontal inflammation: a novel pleiotropic effect of statins. J Am Coll Cardiol. 2013 Dec 24;62(25):2382-2391. doi: 10.1016/j.jacc.2013.08.1627. Epub 2013 Sep 24. PMID 24070911
- [Derived] Tawakol A, Fayad ZA, Mogg R, Alon A, Klimas MT, Dansky H, Subramanian SS, Abdelbaky A, Rudd JH, Farkouh ME, Nunes IO, Beals CR, Shankar SS. Intensification of statin therapy results in a rapid reduction in atherosclerotic inflammation: results of a multicenter fluorodeoxyglucose-positron emission tomography/computed tomography feasibility study. J Am Coll Cardiol. 2013 Sep 3;62(10):909-17. doi: 10.1016/j.jacc.2013.04.066. Epub 2013 May 30. PMID 23727083

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mg Atorvastatin: Participants self-administered one 10 mg atorvastatin tablet and one 80 mg atorvastatin matching placebo tablet orally once daily for 12 weeks.
- 80 mg Atorvastatin: Participants self-administered one 80 mg atorvastatin tablet and one 10 mg atorvastatin matching placebo tablet orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | 10 mg Atorvastatin | 80 mg Atorvastatin
Started | 42 | 41
Completed | 36 | 35
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg Atorvastatin | 80 mg Atorvastatin | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.63) | 59.1 (9.24) | 59.5 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction From Baseline in TBRmeanmax of the Qualifying Segment
Description: Vascular plaque inflammation was measured by 18FDG-PET imaging. Uptake of FDG by the carotid and thoracic aorta is expressed as the target, vessel wall to background, lumen ratio (TBR). TBRmax of an axial cross section of a vessel (a slice) is defined as the maximum TBR within a slice and TBRmeanmax is the mean of TBRmax for all slices in the qualifying segment. The qualifying segment is the left or right carotid or thoracic aorta with the greatest FDG uptake value at Baseline.
Time Frame: Baseline and Week 12
Population: The analysis population includes all participants who completed the study and had complete image sets with usable data.
Measure: Geometric Mean (90% Confidence Interval); unit: Percent reduction
Groups:
- 10 mg Atorvastatin: Participants self-administered one 10 mg atorvastatin tablet and one matching 80 mg atorvastatin placebo tablet orally once daily for 12 weeks.
- 80 mg Atorvastatin: Participants self-administered one 80 mg atorvastatin tablet and one matching 10 mg atorvastatin placebo tablet orally once daily for 12 weeks.
Arm/Group | 10 mg Atorvastatin | 80 mg Atorvastatin
Number analyzed (Participants) | 33 | 34
Percent reduction | 1.4 [-2.6 to 5.3] | 5.8 [2.0 to 9.5]
Statistical Analysis 1: Comparison: 80 mg Atorvastatin; Constrained longitudinal data analysis (cLDA); Test type: Superiority or Other; p = 0.006, cLDA
Statistical Analysis 2: Comparison: 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.277, cLDA
Statistical Analysis 3: Comparison: 10 mg Atorvastatin vs 80 mg Atorvastatin; Test type: Superiority or Other; p = 0.088, cLDA; Percent Reduction = 4.5, 90% CI 2-sided [-1.0 to 9.6]

2. Secondary Outcome: Percent Reduction From Baseline in TBRmeanmax of the Qualifying Segment in Statin-naive Participants
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: The analysis population includes all statin-naive participants who completed the study and had complete image sets.
Measure: Geometric Mean (90% Confidence Interval); unit: Percent reduction
Groups:
- Statin-Naive Participants: Participants self-administered one 10 mg or 80 mg atorvastatin tablet and one matching 80 mg or 10 mg atorvastatin placebo tablet orally once daily for 12 weeks.
Arm/Group | Statin-Naive Participants
Number analyzed (Participants) | 27
Percent reduction | 2.3 [-2.1 to 6.5]
Statistical Analysis 1: Comparison: Statin-Naive Participants; Test type: Superiority or Other; p = 0.195, cLDA

ADVERSE EVENTS:
Arm/Group | 10 mg Atorvastatin | 80 mg Atorvastatin
Serious Adverse Events (participants affected / at risk) | 1/42 | 1/41
Other Adverse Events (participants affected / at risk) | 4/42 | 8/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg Atorvastatin (N=42) | 80 mg Atorvastatin (N=41)
Chest Pain (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg Atorvastatin (N=42) | 80 mg Atorvastatin (N=41)
Alanine Aminotransferase Increased (Investigations) | 1 | 3
Blood Creatinine Phosphokinase Increased (Investigations) | 4 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.